CLINICAL TRIAL: NCT05827003
Title: The Comparison of the Effectiveness of Exercise and Topical Agent Treatments in Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Effects of Exercise Versus Topical Agents on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83483935
Record Dates: First submitted 2023-03-30; First posted 2023-04-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Diclofenac; Non-steroidal anti-inflammatory drugs; Physiotherapy; Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: There will be an equal number of participants in the three groups randomized by the computer.
Who Masked: Investigator
Masking Description: The assessor will not know which participant received which intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise (Active Comparator): Individuals with a diagnosis of knee osteoarthritis who underwent supervised exercise under the guidance of a physiotherapist for 6 weeks, 2 days a week.
  Interventions: Other: Exercise
- Exercise&Topical Agent (Active Comparator): Individuals with a diagnosis of knee osteoarthritis who had supervised exercise under the guidance of a physiotherapist for 6 weeks, 2 days a week, and in addition to this program, they used diclofenac gel 2 times a day, 4 days a week.
  Interventions: Other: Exercise; Other: Exercise&Topical Agent; Other: Topical Agent
- Topical Agent (Active Comparator): Individuals with a diagnosis of knee osteoarthritis using diclofenac gel twice a day, 4 days a week, for 6 weeks
  Interventions: Other: Topical Agent

INTERVENTIONS:
Other: Exercise — Supervised exercise program with a physiotherapist for 6 weeks, two days a week
  Arms: Exercise; Exercise&Topical Agent
Other: Exercise&Topical Agent — Diclofenac gel application to the knee joint twice a day, four days a week, in addition to a supervised exercise program under the supervision of a physiotherapist for 6 weeks.
  Arms: Exercise&Topical Agent
Other: Topical Agent — Application of diclofenac gel to the knee joint twice a day, four days a week, for 6 weeks
  Arms: Exercise&Topical Agent; Topical Agent

SUMMARY:
Osteoarthritis, a chronic and degenerative joint disease, is the most common type of arthritis and affects more than 300 million adults worldwide. Osteoarthritis, which is characterized by joint pain and stiffness, has negative consequences for function, participation and quality of life, which are important components of health. The knee joint is the most common joint in terms of osteoarthritis and is more common in individuals over 50 years of age.

There is no proven definitive treatment in today's literature for common osteoarthritis, which is one of the important causes of the global disease burden. However, since it is a progressive disease with varying degrees of severity, it is a chronic problem that requires long-term treatment. According to current clinical guidelines prepared by the working groups of the International Osteoarthritis Research Society (OARSI) and the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases ESCEO , treatment typically includes physiotherapy interventions with the use of non-steroidal anti-inflammatory drugs (NSAIDs) and analgesics, including intra-articular injections of corticosteroids; In more severe cases, joint replacement surgery is recommended.

The aim of this research project is to examine the effectiveness of a supervised exercise program applied in combination with NSAID-specific topical agents, in comparison with groups receiving only topical agents or only exercise treatments.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with knee osteoarthritis will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into tree groups. Study groups will be as follows: a) exercise, b) exercise & topical agent, c) topical agent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with knee OA according to the criteria of the American Society of Rheumatology
* Stage 2 or 3 according to Kellgren Lawrence radiological staging criteria
* Those between the ages of 40 and 65
* Body mass index below 30 kg/m2
* Pain intensity defined by the patient in the last 3 months is at least 3 out of 10 according to NPRS
* Patients who do not have any obstacles to be included in the exercise program

Exclusion Criteria:

* Using viscosupplementation or steroid injection or systemic steroids in the related knee in the last 3 months
* To have received a physiotherapy program for the relevant knee in the last 3 months
* Having a valgus or varus deformity greater than 15°
* Presence of active infection or tumor
* Presence of neurological diseases and/or deformity leading to lower extremity muscle weakness
* Having serious systemic and cardiovascular diseases that interfere with exercise

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change of Pain via Numeric Pain Rating Scale | change from baseline pain at 6 months
  On this scale, "0" indicates the absence of pain, and "10" indicates the most severe pain imaginable (17). Patients will be asked to rate the severity of their knee pain with a number between 0 and 10 using this scale. The minimum clinically significant difference value (MCID) of this valid and reliable pain scale is 1.74 points.

SECONDARY OUTCOMES:
WOMAC | 4 times for 24 weeks
  WOMAC assesses the level of difficulty, pain and joint stiffness experienced by the patients during their physical functions. WOMAC score is a 5-point Likert-type scale, high scores indicate poor status and consist of a total of 24 questions.
40 meters fast walking test | 4 times for 24 weeks
  For 40mHYT, patients will be asked to walk as fast as possible on a flat and hard surface, on a 10-meter marked walking path. Walking time will be measured in seconds with a stopwatch. The test will be repeated three times and the arithmetic mean of these measurements will be recorded as the result value. Considering the age range of the patients, it was planned to allow a one-minute rest period between retests.
Stepping Test | 4 times for 24 weeks
  Patients will be asked to climb 10 pre-marked 20 cm high steps as quickly as possible on a standard ladder. The test time will be measured in seconds with a stopwatch. The test will be repeated 3 times and the average value will be recorded in seconds. Similarly, in this evaluation, patients were given a one-minute rest period between 3 repetitions of the test.
Joint Range of Motion Evaluation | 4 times for 24 weeks
  During the assessments, three repeat measurements will be made using an electronic goniometer. For goniometric measurement, the pivot point will be placed on the lateral condyle of the femur. The fixed arm will be held parallel to the lateral midline of the femur. The movable arm will follow the movement of the fibula.
Health-Related Quality of Life Short Form (SF-12) Scale | 4 times for 24 weeks
  SF-12 is the abbreviated version of the SF36 Quality of Life Scale and is frequently preferred for ease of use. It has 2 components, physical and mental, scored between 0 and 50.
  A high score from the score indicates health-related well-being and increased quality of life, while a decrease indicates worsening.
Global Rating of Change Scale-GRC | 3 times for 24 weeks
  It will be used to evaluate patient satisfaction. It is designed to determine the amount of improvement or worsening of the patient over time.
  In our study, GRC consisting of 5 levels between -2 and +2 value ranges (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) was preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Celik, Prof., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Safiri S, Kolahi AA, Smith E, Hill C, Bettampadi D, Mansournia MA, Hoy D, Ashrafi-Asgarabad A, Sepidarkish M, Almasi-Hashiani A, Collins G, Kaufman J, Qorbani M, Moradi-Lakeh M, Woolf AD, Guillemin F, March L, Cross M. Global, regional and national burden of osteoarthritis 1990-2017: a systematic analysis of the Global Burden of Disease Study 2017. Ann Rheum Dis. 2020 Jun;79(6):819-828. doi: 10.1136/annrheumdis-2019-216515. Epub 2020 May 12. PMID 32398285
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] Bruyere O, Honvo G, Veronese N, Arden NK, Branco J, Curtis EM, Al-Daghri NM, Herrero-Beaumont G, Martel-Pelletier J, Pelletier JP, Rannou F, Rizzoli R, Roth R, Uebelhart D, Cooper C, Reginster JY. An updated algorithm recommendation for the management of knee osteoarthritis from the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Semin Arthritis Rheum. 2019 Dec;49(3):337-350. doi: 10.1016/j.semarthrit.2019.04.008. Epub 2019 Apr 30. PMID 31126594
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Gregori D, Giacovelli G, Minto C, Barbetta B, Gualtieri F, Azzolina D, Vaghi P, Rovati LC. Association of Pharmacological Treatments With Long-term Pain Control in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. JAMA. 2018 Dec 25;320(24):2564-2579. doi: 10.1001/jama.2018.19319. PMID 30575881
- [Background] Arden NK, Perry TA, Bannuru RR, Bruyere O, Cooper C, Haugen IK, Hochberg MC, McAlindon TE, Mobasheri A, Reginster JY. Non-surgical management of knee osteoarthritis: comparison of ESCEO and OARSI 2019 guidelines. Nat Rev Rheumatol. 2021 Jan;17(1):59-66. doi: 10.1038/s41584-020-00523-9. Epub 2020 Oct 28. PMID 33116279
- [Background] van Doormaal MCM, Meerhoff GA, Vliet Vlieland TPM, Peter WF. A clinical practice guideline for physical therapy in patients with hip or knee osteoarthritis. Musculoskeletal Care. 2020 Dec;18(4):575-595. doi: 10.1002/msc.1492. Epub 2020 Jul 9. PMID 32643252
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142